CLINICAL TRIAL: NCT01086345
Title: Phase I/II Trial of Radiosurgery Plus Bevacizumab in Patients With Recurrent/Progressive Glioblastoma
Brief Title: Radiosurgery Plus Bevacizumab in Glioblastoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4309; NCI-2010-00309 (Other: NCI/CTRP)
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Glioblastoma; Gliosarcoma; Brain Tumor
Keywords: adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Radiosurgery; Bevacizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive bevacizumab IV over 30 minutes on days 1 and 15. Patients also receive irinotecan hydrochloride IV on days 1 and 15 beginning in course 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo radiosurgery 10-14 days after beginning bevacizumab.
  Interventions: Radiation: radiosurgery; Biological: bevacizumab; Drug: irinotecan hydrochloride

INTERVENTIONS:
Radiation: radiosurgery — Patients undergo radiosurgery 10-14 days after beginning bevacizumab.
  Other Names: Radiation Surgery
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; Avastin; recombinant humanized anti-VEGF monoclonal antibody; rhuMAb VEGF
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; camptothecin-11; CPT-11; irinotecan; U-101440E

SUMMARY:
RATIONALE: Radiosurgery can send x-rays directly to the tumor and cause less damage to normal tissue. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of glioblastoma by blocking blood flow to the tumor. Drugs used in chemotherapy such as irinotecan hydrochloride work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiosurgery together with bevacizumab and irinotecan hydrochloride may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving radiosurgery together with bevacizumab and irinotecan hydrochloride works in treating patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall survival of patients with recurrent GBM treated with bevacizumab, irinotecan and radiosurgery

SECONDARY OBJECTIVES:

I. To evaluate the toxicities of the combination of bevacizumab, irinotecan and radiosurgery.

II. To evaluate the progression-free survival of patients treated with bevacizumab, irinotecan and radiosurgery.

OUTLINE:

Patients receive bevacizumab IV over 30 minutes on days 1 and 15. Patients also receive irinotecan hydrochloride IV on days 1 and 15 beginning in course 2. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo radiosurgery 10-14 days after beginning bevacizumab.

After completion of study treatment, patients are followed for 18 months.

ELIGIBILITY:
Inclusion

* Histologically proven diagnosis of glioblastoma or gliosarcoma (WHO grade IV) at primary or subsequent resection
* Radiographic evidence of tumor progression as defined by a contrast enhanced MRI at least 3 months after the completion of radiation therapy
* Unifocal enhancing disease; the enhancing focus must be =< 3 cm in maximum diameter
* History/physical examination within 14 days prior to registration
* The patient must have recovered from the effects of prior therapy before study entry
* The patient must not have received chemotherapy within the following time frames: Non-cytotoxic agents: 2 weeks, cytotoxic agents: 3 weeks, nitrosoureas: 6 weeks
* Must be able to undergo MRI imaging
* Documentation of steroid doses within 14 days prior to registration
* Karnofsky performance status > 60
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 10.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb >= 10.0 g/dl is acceptable)
* BUN =< 30 mg/dl within 14 days prior to study entry
* Creatinine =< 1.7 mg/dl within 14 days prior to study entry
* Urine protein screened by urine analysis for urine protein creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg
* Bilirubin =< 2.0 mg/dl within 14 days prior to study entry
* ALT/AST =< 3 x normal range within 14 days prior to study entry
* Electrocardiogram without evidence of acute cardiac ischemia within 14 days prior study entry
* Prothrombin time/international normalized ratio (PT INR) < 1.4 for patients not on warfarin confirmed by testing within 14 days prior to study entry
* Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria: No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices); in-range INR (between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
* Patients must provide study specific informed consent prior to study entry
* Women of childbearing potential and male participants must practice adequate contraception
* For females of child-bearing potential, negative serum pregnancy test within 14 days prior to entry

Exclusion

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for >= 3 years (for example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible)
* More than one focus of enhancement
* Involvement of the brainstem (defined as the midbrain or lower)
* Prior use of chemotherapy wafers or any other intratumoral or intracavitary treatment are not permitted; prior radiosurgery is not permitted
* Prior treatment with intravenous bevacizumab
* Unstable angina and/or congestive heart failure within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an EKG performed within 14 days of entry
* New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration
* History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months
* Serious and inadequately controlled cardiac arrhythmia
* Uncontrolled hypertension
* Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for tumor resection
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of entry
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of entry
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
* Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol
* Active connective tissue disorders, such as lupus or scleroderma that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study drug
* Patients treated on any other therapeutic clinical trials within 30 days prior to study entry or during participation in the study
* Growth factors are not permitted to induce elevations in neutrophil count for the purposes of: 1) administration of temozolomide on the scheduled dosing interval; 2) allowing treatment with temozolomide at a higher dose; or 3) avoiding interruption of the treatment during concomitant radiotherapy
* No other investigational drugs will be allowed during this study
* Surgical procedures for tumor debulking, other types of chemotherapy, and immunotherapy or biologic therapy must not be used
* Additional stereotactic boost radiotherapy is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall survival of patients with recurrent GBM treated with bevacizumab, irinotecan and radiosurgery | Patients are followed for 18 months.

SECONDARY OUTCOMES:
Treatment-related toxicity | Courses repeat every 28 days in the absence of unacceptable toxicity.
Progression-free survival, defined as the interval from randomization to progression or death, whichever occurs first | Patients are followed for 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vogelbaum, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States